CLINICAL TRIAL: NCT06512623
Title: Cytokine Adsorption During Complex Cardiac Surgery: the JACCS Controlled Randomized Clinical Trial
Brief Title: Cytokine Adsorption During Complex Cardiac Surgery: a Controlled Randomized Trial
Acronym: JACCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Antoine Schneider, Principal Investigator, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CER-VD-2024-D0057
Record Dates: First submitted 2024-07-01; First posted 2024-07-22 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Post-cardiac Surgery; Inflammation; Organ Dysfunction Syndrome; Cardiac Disease; Cardio-Pulmonary Bypass
Keywords: Post-pump syndrom; Cytokine Hemoadsorption; Post-operative organ failure
MeSH Terms: conditions — Inflammation; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Cardiopulmonary bypass will be conducted as per institutional protocols, without hemoadsorption (standard-of-care)
- Hemoadsorption (Experimental): Cardiopulmonary bypass (CPB) will be conducted as per institutional protocols and an HA-380® cartridge (Jafron Biomedical, Guangdong, China) will be inserted within the circuit for hemoadsorption.
  Interventions: Device: Hemoadsoprtion

INTERVENTIONS:
Device: Hemoadsoprtion — The hemoadsorption treatment will be performed during the entire duration of the CPB. Blood flow within the cartridge is standardized at 250 ml/min.
  Arms: Hemoadsorption

SUMMARY:
This prospective single-centre randomized controlled trial aims at evaluating the safety and efficacy of hemoadsorption with HA-380® during cardio-pulmonary bypass in 40 patients undergoing complex cardiac surgery.

DETAILED DESCRIPTION:
Cardiopulmonary bypass (CPB) is an extracorporeal circuit used to divert blood from the heart and lungs and take over their functions during cardiac surgery. Cardiac surgery with CPB can induce a major inflammatory response, largely mediated by cytokines. In the most severe cases, this inflammation can lead to vasoplegia, hypotension and potentially end-organ damage.

The investigators hypothesised that the removal of inflammatory mediators (e.g. cytokines) from the blood during CPB could reduce the development of postoperative complications in patients with significant inflammation during cardiac surgery.

Patients undergoing complex cardiac surgery will be enrolled preoperatively and randomised 1:1 to receive either the investigational hemoadsorption treatment plus standard care (intervention group) or standard care alone (control group). Patients allocated to the intervention group will have an HA-380® cartridge (Jafron Biomedical, Guangdong, China) inserted into the CPB during circuit set-up. Hemoadsorption treatment will be performed throughout the duration of the CPB procedure.

For each patient, 4 blood samples will be taken for cytokine measurements (at the start of CPB, at the end of CPB, at ICU admission and 24 hours later). Data on vital signs, organs support, demographics and medical history will be collected in the electronic medical record.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥18 years old at study inclusion)
2. Planned for one of the following cardiac surgical procedures: heart transplantation after L-VAD (left ventricular assist device) implantation, OR surgical repair of a type A aortic dissection, OR urgent (within a few days) or emergent (within 24 hours) procedure for acute infectious endocarditis, OR cardiac surgery likely to require >180 min CPB time as estimated by the surgical team
3. Signed informed consent

Exclusion Criteria:

1. Indication to receive hemoadsorption during CPB for drugs removal
2. Women who are pregnant or breastfeeding
3. Previous enrolment into the current study
4. Off-pump procedure
5. Chronic immunosuppression
6. Known allergy to heparin or heparin induced thrombocytopenia
7. Severe thrombopenia (platelets count before surgery < 20g/L)
8. Patient who does not want to be informed of incidental findings
9. Participation in another study with investigational drug within the 30 days preceding and during the present study
10. Participation in another conflicting research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2024-10-27 (Actual); Primary Completion 2025-12-18 (Actual); Study Completion 2026-01-12 (Actual)

PRIMARY OUTCOMES:
SOFA score at 24 hours | Within 24 hours of ICU admission
  Difference between groups in the SOFA score measured within 24 hours after ICU admission

SECONDARY OUTCOMES:
ICU and hospital length of stay | At time of hospital discharge, an average 20 days after ICU admission
  Lengths of stays, in days
ICU, hospital, and 28 days (from ICU admission) mortality | At time of hospital discharge, an average 20 days after ICU admission and up to 28 days after ICU admission
  All-cause mortality
Days alive without respiratory support | At day 28 from ICU admission
  Number of days alive and without mechanical ventilation
Days alive without renal replacement therapy | At day 28 from ICU admission
  Number of days alive and without renal replacement therapy
Days alive without vasopressors | At day 28 from ICU admission
  Number of days alive and without vasopressors
SOFA score at 48 hours | Measured between 24 hours and 48 hours after ICU admission
  Sequential Organ Failure Assessment (SOFA) difference between groups in the SOFA score measured between 24hours and 48 hours after ICU admission. The higher the SOFA the highest the probability of death
Post-operative complications | At time of ICU discharge, up to 7 days after ICU admission
  Post-operative Acute Kidney Injury, transfusion of red blood cells, sepsis, delirium, liver injury or need for coronary angiography
Cytokines levels | at the end of CPB, at the admission in ICU and 24 hours after ICU admission
  Relative and absolute reduction in the plasma levels of cytokines at different timepoints, compared with their levels at baseline (immediately before CPB initiation).

OTHER OUTCOMES:
Device-related complications | During cardiopulmonary bypass
  Technical failure to perform the treatment (thrombosis of cartridge, circuit leak, inability to perform the treatment for all CPB duration)
Treatment tolerance | During cardiopulmonary bypass
  New allergic or anaphylactoid reaction (stage ≥ 2 according to H. L. Mueller [39]) or new fever (> 38.5°C)
Safety of intervention | From beginning of cardiopulmonary bypass to 7 days after ICU admission,
  Bleeding and haematological complications Post-operative infections New acute organ rejection
Feasibility of intervention | During cardiopulmonary bypass
  Screened to enrolled patients' ratio, success of intervention delivery in intervention group, duration of recruitment

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Schneider, Principal Investigator — CHUV Centre Hospitalier Universitaire Vaudois (CHUV)
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No